CLINICAL TRIAL: NCT02655965
Title: A Randomised, Double-blind, Placebo-controlled Study to Assess the effectIveness of Pectoral Nerves Block (PECS) After Breast Surgery on Piritramide Consumption
Brief Title: Double-blind Study to Assess effectIveness of Pectoral Nerves Block After Breast Surgery on Piritramide Consumption
Acronym: DESIGN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IJB-SUR-DESIGN-2015; 2015-005574-38 (EudraCT Number); CE2483 (Other: Institut Jules Bordet)
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Locoregional Analgesia in Breast Surgery
Keywords: Breast cancer; lumpectomy; mastectomy; PECS bloc
MeSH Terms: conditions — Breast Neoplasms | interventions — Ropivacaine; Clonidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine + Clonidine (Experimental): A "pecs block" of Ropivacaine 3.5 mg/ml and Clonidine 5 µg/ml will be injected to the patients prior surgery. 10 ml of the drug combination will be injected between pectoral muscles and 20 ml of the drug combination will be injected between the muscles pectoralis minor and serratus anterior.
  After surgery, subjects in both arms will receive one dose of Paracetamol (1g) and Diclofenac (75 mg) and one dose 0.05 mg/kg Piritramide as well as PCIA (Patient Controlled Intravenous Analgesia)-Piritramide for 24 hrs post-surgery.
  Interventions: Drug: Ropivacaine; Drug: Clonidine
- Sodium Chloride (Placebo Comparator): A "pecs block" of Placebo (Sodium Chloride 0.9%) will be injected to the patients prior surgery. 10 ml of the Sodium chloride solution will be injected between pectoral muscles and 20 ml of the Sodium chloride solution will be injected between the muscles pectoralis minor and serratus anterior).
  After surgery, subjects in both arms will receive one dose of Paracetamol (1g) and Diclofenac (75 mg) and one dose 0.05 mg/kg Piritramide as well as PCIA (Patient Controlled Intravenous Analgesia)-Piritramide for 24 hrs post-surgery.
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine 3.5 mg/ml
  Arms: Ropivacaine + Clonidine
Drug: Clonidine — Clonidine 5µg/ml
  Arms: Ropivacaine + Clonidine
Drug: Sodium Chloride — Sodium Chloride 0.9 %
  Arms: Sodium Chloride

SUMMARY:
The aims of this study is to compare the effectiveness of pecs block associated to a general anesthesia in terms of Piritramide consumption compared with a general anaesthesia alone and the chronic pain incidence in patients that undergoing either a lumpectomy or a mastectomy associated with axillary dissection This is a double-blind, placebo controlled study that will randomise breast cancer subjects in 1:1 ratio to receive a "pecs block" of Ropivacaine 3.5 mg/ml and Clonidine 5 µg/ml (arm A) versus placebo (arm B).

DETAILED DESCRIPTION:
This is a double-blind study that will randomise breast cancer subjects in 1:1 ratio to receive a "pecs block" of 10 ml of Ropivacaine 3.5 mg/ml and Clonidine 5 µg/ml injected between pectoral muscles and 20 ml between the muscles pectoralis minor and serratus anterior (arm A) versus 10 ml of placebo (NaCl 0.9%) injected between pectoral muscles and 20 ml between the muscles pectoralis minor and serratus anterior (arm B). The pecs block will inject just before the surgery.

Subjects will receive a nausea and vomiting prophylaxy depending on Apfel score After surgery, the two intervention groups will receive before waking a dose of Paracetamol (1 g) and Diclofenac (75 mg), if they present no contraindications and a dose of 0.05 mg/kg Piritramide .

In the recovery room the two groups will benefit from a Patient Controlled Intravenous Analgesia (PCIA) pump - Piritramide allowing them to control their analgesia, which will be stopped at 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Female
3. Subjects undergoing either a conservative or non-conservative breast surgery associated with axillary dissection
4. ASA score ≤ 3
5. Completion of all necessary screening procedures within 30 days prior to randomisation
6. Adequate Renal Function including: Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥ 60 ml/min as calculated using the method standard for the institution
7. Adequate Liver Function, including all of the following parameters:

   1. Aspartate and Alanine Aminotransferase (AST and ALT) ≤ 1.5 x ULN If Aspartate and Alanine aminotransferase (AST and ALT) are > 1.5 x ULN, total serum bilirubin should be assessed and must be ≤ 1.5 x ULN unless the patient has documented Gilbert Syndrome
   2. Alkaline phosphatase ≤ 2.5 x ULN
8. Signed informed consent
9. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures

Exclusion criteria:

1. Any illness or medical condition that is unstable or could jeopardize the safety of the patient or her compliance with study requirements
2. Allergy to local anaesthetics
3. Known allergy or hypersensitivity to Paracetamol, Diclofenac, Piritramide or excipients
4. Coagulopathy or taking oral anticoagulant/ antiaggregant within 7 days prior to surgery
5. BMI> 35 kg / m2
6. Infection near the puncture site
7. Inability to understand the pain assessment scales (VAS and McGill questionnaire)
8. Severe hepatic impairment: elevated transaminases with factor V ≤ 50%
9. Severe heart failure: NYHA classification III or IV and/or LVEF < 50%
10. Pregnant or lactating women
11. Concurrent treatment with daily basis chronic opiate type painkillers not ended 1 month prior surgery
12. Scheduled breast reconstruction at the time of surgery
13. Metastatic subjects
14. Subjects with breast implants
15. Patients that require bilateral mastectomy or bilateral lumpectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-05; Primary Completion 2019-11 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of pecs block in terms of total Piritramide consumption | 24 hrs post-surgery
  Piritramide consumption in the first 24 h post-surgery will be recorded

SECONDARY OUTCOMES:
Evaluation of incidence of chronic pain in both groups at 6 months postoperatively | 6 months post-surgery
  Pain intensity until 6 months post-surgery will be evaluated using the Short version of Mc Gill questionnaire (SF-MPQ2)
Evaluation of present pain post-operatively | 48 hours post-surgery
  Present pain intensity until 48 hrs post- surgery will be assessed by Visual Analog scoring

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Sosnowski, MD, Study Chair — Jules Bordet Institute; Kathleen Wiams, MD, Study Chair — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No